CLINICAL TRIAL: NCT06075485
Title: Management of Drug-resistant Epilepsy in Infants and Children: a Real-life Study of the Use of the Ketogenic Diet in France and the KetoCal® Range in Its Maintenance
Acronym: KEOPS
Status: Recruiting | Type: Observational
Sponsor: Nutricia Nutrition Clinique (Industry)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A01073-42
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Drug Resistant Epilepsy; Ketogenic Dieting
Keywords: ketogenic diet; epilepsy; drug resistance
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Infants (from 5 months) and children up to 17 years of age follow up for drug resistant epilepsy
  Interventions: Other: Ketocal

INTERVENTIONS:
Other: Ketocal — ketogene diet

SUMMARY:
This is a multicenter, prospective, observational, longitudinal study designed to describe the therapeutic value of the KetoCal® range in the maintenance of a ketogenic diet during the management of infants (from 5 months) and children up to 17 years of age (i.e. 18 years minus 1 day) with drug-resistant epilepsy.

This study is being conducted according to standard medical practice. No change in diagnostic or therapeutic management habits is imposed by this study. Quality of life questionnaires are the only additional procedures for this research.

DETAILED DESCRIPTION:
NUTRICIA has developed the KetoCal® range (4:1 and 3:1), a food for special medical purposes (DADFMS), to help healthcare professionals and patients establish and maintain a CR. KetoCal® 4:1 features a 4:1 ratio of fat to (carbohydrate + protein), while containing vitamins, minerals, trace elements and fiber. Similarly, KetoCal® 3:1 has a 3:1 ratio of lipids / (carbohydrates + proteins), while containing vitamins, minerals, trace elements and fiber. The KetoCal® range can be consumed orally, as a drink after dilution in hot water, incorporated as an ingredient in a recipe or administered by enteral feeding tube.

The KEOPS study is designed to gather real-life data on the therapeutic value of using the KetoCal® range in the management of drug-resistant epilepsy in infants (from 5 months) and children up to 18 years of age. Patients will be managed according to standard care practices. Initiation of ketogenic dieting will be at the investigator's discretion during the child's hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Infants from 5 months and children up to 17 years of age (maximum 18 years minus 1 day).
* With drug-resistant epilepsy according to ILAE (International League Against Epilepsy) criteria: persistence of epileptic seizures after failure of two appropriate antiepileptic drugs tried consecutively or in well-tolerated combination.
* Indication for CR by a physician.
* Parents (or legal guardians) able to set up and follow the diet, assessed during a joint doctor-dietician consultation.
* Written authorization from one (or both) parents or the child's legal representative to collect personal information about their child.
* Affiliation of the infant/child with the social security system.

Exclusion Criteria:

* Contraindication to ketogenic diet at initial assessment.
* Children already on a ketogenic diet.
* Parenteral nutrition.
* Concurrent prescription of other foodstuffs intended for special medical purposes (DADFMS) such as KetoVie or Keyo.
* Protected legal representative (under legal protection, or deprived of liberty by judicial or administrative decision).
* Legal representative not covered by a social security scheme.
* Legal representative unable to understand study protocol.

Ancillary study eligibility criteria :

* Patients included in the study.
* Continued on the ketogenic diet for at least 2 months.
* Having consented to participate in the ancillary study.

Ages: 5 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 133 eligible patients will be recruited in this project. The target population of our project will be infants (from 5 months of age) and children up to 18 years of age treated for drug-resistant epilepsy, who, depending on the physician in charge of the patient, may benefit from the initiation of a KetoCal® 3:1 or 4:1 CR, depending on the child's age.
  We exclude from our study protected legal representatives of minors (under guardianship, curatorship, minor parents). In addition, people taking part in this study will not be able to take part in any other interventional or observational research for the duration of the study. A 6-month exclusion period is planned as part of this project.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Description of compliance | 6 months
  Retention rate which is defined as the proportion of patients who have continued KD for up to 6 months.

SECONDARY OUTCOMES:
Duration of compliance | From Month 1 to Month 6
  Describe the duration of KD compliance.
Efficacy of KD | From Month 1 to Month 6
  Describe the efficacy of KD. Efficacy is defined as responders to KD with seizure frequency reduced by more than 50%, or no seizure frequency in the case of total response to CR in the last week.
KD tolerance. | From inclusion to Month 6
  Describe KD tolerance as a number of AE reported
QoL evolution | From inclusion to Month 6
  Describe changes in patients' quality of life following initiation of KD at inclusion, and M6; using PedsQL ™ questionnaires
Influence of KD | From inclusion to Month 6
  Total number of antiepileptic drugs used for each child including their current treatment until the end of the study.
Ketosis achievement | From inclusion to Month 6
  Evaluate the time it takes to achieve ketosis. Ketosis will be assessed by ketonuria or ketonemia, depending on the habits of each center.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No